CLINICAL TRIAL: NCT02542917
Title: Home Versus Postal Testing for Faecal Calprotectin: a Feasibility Study
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15/WA/0518
Record Dates: First submitted 2015-05-29; First posted 2015-09-07 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: IBDoc home test for faecal calprotectin
  Interventions: Device: IBDoc home test for faecal calprotectin

INTERVENTIONS:
Device: IBDoc home test for faecal calprotectin — IBDoc home test for faecal calprotectin

SUMMARY:
This trial will test, in a representative group of IBD patients, the acceptability of - and adherence to - the IBDoc test (a new home test for faecal calprotectin in the monitoring of inflammatory bowel disease (IBD)).

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are forms of inflammatory bowel disease (IBD) that require long-term monitoring. People with these conditions require regular and repeat testing, sometimes with endoscopy, to assess the state of the disease. Many centres worldwide now use a stool test called faecal calprotectin (FCALP) as an accurate reflection of endoscopic disease activity - meaning that people with IBD do not need 'routine' endoscopy to assess their disease. FCALP can also be used to give a prediction of what will happen to a person's IBD in the near future.

As such, FCALP is an excellent and highly cost-effective test in IBD. However, uptake is often low (as with all stool tests) particularly because the sample needs to be taken at home and delivered in to the laboratory or hospital to be tested. People still therefore need to make an effort to submit samples and find this inconvenient. Furthermore, treatments for IBD are increasingly being given at home (usually self-administered injections). While beneficial for people with IBD, it is more difficult to keep track of such patients in the hospital service as they attend less regularly. A test that can be done at home, while making results available to the hospital team, is therefore desirable.

New technology allows reliable testing of FCALP at home, using a smartphone app (IBDoc-TM, Buhlmann Laboratories) within a few minutes. The test kit is packaged with everything required (including gloves, sample 'capture' paper, disposal bag, etc). An instructional video is available within the app itself.

Apart from testing whether patients adhere to the testing schedule, the investigators will also compare their experiences of the IBDoc test, health anxieties, locus of control, and satisfaction vs postal and traditional 'drop-off' test. Validated questionnaires will include: GAD7, PHQ9, IBDC, CBRQ and MHLC as well as a proprietary satisfaction questionnaire at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease diagnosed at least 6 months prior to study entry
* Willing to participate in home testing and have smartphone
* Able to understand English or explanation via interpreter, and provide written consent

Exclusion Criteria:

* Participants without smartphone (Android or iOS)
* Unable to understand English (excl. via interpreter)
* No previous experience of submitting stool samples for faecal calprotectin measurement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected patients with any form of inflammatory bowel disease on any treatment and at any stage of disease activity (diagnosed more than 6 months prior to study entry)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Adherence to testing schedule (overall >75%) | 6 months
  As this is a feasibility study there is no 'outcome' measure as such; We are testing the adherence to the study protocol as the main outcome of this study

SECONDARY OUTCOMES:
Any change in health locus of control score | 6 months
  Any change in MHLC score from study start to end
Any change in cognitive behavioural response score | 6 months
  Any change in CBRQ-32 score from study start to end

CONTACTS AND LOCATIONS:
Overall Officials: Bu'Hussain Hayee, Principal Investigator — King's College Hospital NHS Trust